CLINICAL TRIAL: NCT02375438
Title: Nutritional Assessment in Patients Affected by Mitochondrial Cytopathy
Brief Title: Nutritional Assessment in Mitochondrial Cytopathy
Acronym: NAMITO
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 242/14; Insel 2660 (Other: University hospital Berne); KEK 242/14 (Other: Ethics Committee)
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Cytopathies
Keywords: nutrition; mitochondrial cytopathy; malnutrition; energy intake; nutritional risk
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial cytopathy; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine. All samples collected in this study (blood and urinary) will be sent to a central biobank for long term storage.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort Group: Patients with a clinical presentation suggestive of mitochondrial cytopathy, in whom mitochondrial deletions above 20% have been found in muscle are considered eligible if they are older than 18 years and are willing and able to give written informed consent.
- Control Group: Twenty healthy individuals matched for age and gender will be included in the study and considered as controls.

SUMMARY:
The aim of this study is to assess nutritional intake (quantitatively and qualitatively), nutritional state and body composition of patients suffering from mitochondrial cytopathy, compared to healthy controls. The energy intake will be calculated through dietary protocols, the energy expenditure by indirect calorimetry and body composition will be performed with bio-impedance analysis. Further on, the investigators expect to be able to provide nutritional counselling to this population in order to increase energy and protein intake, which may improve health and well-being.

DETAILED DESCRIPTION:
Background

Mitochondrial diseases are a group of genetic disorders. The prognosis for patients with mitochondrial myopathies varies greatly, depending largely on the type of disease and the degree of involvement of various organs. This situation can lead into malnutrition and worse the outcome. In the literature there are no data, which deal with malnutrition or nutritional intake in patients with mitochondrial myopathy. Sorensen et al. assessed the malnutrition risk in European hospitals and showed that 45% of patients with neurological illness (neurological vascular disease excluded) are at high risk of malnutrition. Furthermore, the patient at risk exhibited higher rates of complications and mortality. These findings suggest that malnutrition play an important role in the clinical outcome of this patient's population, reflecting the investigators' many years of experience. In several case reports, it was shown that malnutrition itself could aggravate myopathy. Sometimes there are challenging symptoms facing patients with mitochondrial myopathy that interfere with obtaining balanced and healthy nutrition, such as fatigue, muscle weakness, dysmotility, dysphagia, nausea and vomiting, ataxia, and reflux. In addition, in the investigators' clinical experience, they see many patients who describe that some specific food intake would even modify their symptoms.

This is an observational cohort study, and the investigators expect a total sample size of 30 patients and 20 healthy age- and sex-matched controls. The entire study will be conducted during the period from first of October 2014 till End of March 2015.

The investigator is a pharmacy student (master level) interested in clinical nutrition. She will collect the data und do all measurements along with the support of the clinical nutrition research team of the University Hospital of Bern. The investigator will contact the patients individually and arrange a suitable timetable for the interview and examination. Sex, age, current medical conditions, current myopathy symptoms, current gastrointestinal symptoms, unintentional weight loss, eating and drinking habits, living and social situation, daily activity, medications (in particular those drugs that interfere with the mitochondrial metabolism as valproic acid, statins, and certain antibiotics like aminoglycosides, etc.) smoking, alcohol intake, and main diagnosis will be recorded. The investigators will preform the following measurements: basic demographic data, structured patient interviews, dietary questionnaire, nutritional risk screening, quality of life, physical functioning, body composition, energy expenditure, blood and urine analysis. The study will be conducted in accordance with the ethical guidelines of the 1957 Declaration of Helsinki, and informed consent will be obtained from all participants. The healthy volunteers and patients will not be exposed to any risk due to this study.

Objective

The aim of this study is to assess the nutritional intake and the nutritional state of patients with mitochondrial myopathy compared to healthy controls. The investigators expect to be able to provide general nutritional advice (nutritional counselling) to increase the ingestion of balanced/healthy food and the energy intake, and therefore they expect to improve health and well-being in this population.

Methods

Questionnaire, indirect calorimetry, bioimpedance analysis BIA, Hand grip test, Anthropometrics and 7-days food recall protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical presentation suggestive of mitochondrial cytopathy, in whom mitochondrial deletions above 20% have been found in muscle
* =/>18 years
* Willing and able to give written informed consent

Exclusion Criteria

* Patients with poor knowledge of the study languages (German and French)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients affected by mitochondrial cytopathy from the outpatient's clinic of the Department of Neurology of the University Hospital of Bern who fulfill the inclusion criteria will be asked to participate in the study. All potential participants will be provided with a patient information sheet and will be given adequate time to consider participation in the study. Those who will participate will be asked to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Energy and nutrients intake (Measured in kcal) | At baseline
  Measured in kcal (7 days food recall protocol to check for nutrients which aggravate symptoms & to provide nutritional counselling)

SECONDARY OUTCOMES:
Differences in nutritional risk (Measured in NRS2002) | At baseline
  Measured in NRS2002 score points
Differences in nutritional status Measured in laboratory parameters (blood and urine) | At baseline
  Measured in laboratory parameters (blood and urine)
Difference in body composition Measured in bioimpedance analysis BIA and anthropometrics (TSF [mm], MAMC (cm^2), Handgrip test (kg)) | At baseline
Difference in resting energy expenditure Measured in kcal (indirect calorimetry) | At baseline
  Measured in kcal (indirect calorimetry)
Difference in quality of life Measured in SF36v2 score | At baseline
  Measured in SF36v2 score

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Stanga, Prof. Dr. med. MD, Principal Investigator — Department of Endocrinology, Diabetes and Clinical Nutrition University Hospital
Locations (1):
- Department of Endocrinology, Diabetes and Clinical Nutrition, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Arpa J, Cruz-Martinez A, Campos Y, Gutierrez-Molina M, Garcia-Rio F, Perez-Conde C, Martin MA, Rubio JC, Del Hoyo P, Arpa-Fernandez A, Arenas J. Prevalence and progression of mitochondrial diseases: a study of 50 patients. Muscle Nerve. 2003 Dec;28(6):690-5. doi: 10.1002/mus.10507. PMID 14639582
- [Background] El-Hattab AW, Scaglia F. Mitochondrial DNA depletion syndromes: review and updates of genetic basis, manifestations, and therapeutic options. Neurotherapeutics. 2013 Apr;10(2):186-98. doi: 10.1007/s13311-013-0177-6. PMID 23385875
- [Background] Sorensen J, Kondrup J, Prokopowicz J, Schiesser M, Krahenbuhl L, Meier R, Liberda M; EuroOOPS study group. EuroOOPS: an international, multicentre study to implement nutritional risk screening and evaluate clinical outcome. Clin Nutr. 2008 Jun;27(3):340-9. doi: 10.1016/j.clnu.2008.03.012. Epub 2008 May 27. PMID 18504063
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673